CLINICAL TRIAL: NCT03287674
Title: T-cell Therapy in Combination With Checkpoint Inhibitors for Patients With Advanced Ovarian-, Fallopian Tube- and Primary Peritoneal Cancer
Brief Title: TIL Therapy in Combination With Checkpoint Inhibitors for Metastatic Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, M.D., Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GY1721
Record Dates: First submitted 2017-09-14; First posted 2017-09-19 (Actual); Results first posted 2021-03-22 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Interleukin-2; Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient group (Experimental): All patients receive the same treatment. All patients are treated with one dose of Ipilimumab 14 days prior to surgical removal of tumor tissue for TIL expansion. Hospitalization for TIL treatment is approximately 3 weeks.
  The patients are admitted to hospital on day -8 and receive lymphodepleting chemotherapy (cyclophosphamide and fludarabine= on day -7 to day -1. The first of 4 doses of Nivolumab is administered on day -2 and every 2 weeks for at total of 4 doses.
  The TILs are infused on day 0 and Interleukin-2 therapy is administered on day 0 to day 13.
  Interleukin-2 is administered as a daily low-dose subcutaneous injection for a total for 14 days.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: TIL infusion; Drug: Interleukin-2; Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 60 mg/kg is administered i.v. on day -7 and day -6.
Drug: Fludarabine — Fludarabine 25 mg/m2 is administered on day -5 to day -1.
  Other Names: Fludarabine phosphate
Biological: TIL infusion — The maximum number of expanded TILs are infused over 30-45 minutes on day 0.
  Other Names: TILs
Drug: Interleukin-2 — Interleukin-2 is administered as a daily low-dose subcutaneous injection of 2 MIU for a total of 14 days.
  Other Names: IL-2
Drug: Ipilimumab — One dose of Ipilimumab 3 mg/kg is administered 14 days prior to surgical removal of tumor tissue for TIL expansion.
Drug: Nivolumab — Nivolumab 3 mg/kg is administered on day -2 before TIL infusion and every 2 weeks for a total of 4 doses.

SUMMARY:
Adoptive T cell therapy (ACT) with tumor infiltrating lymphocytes (TIL) has achieved impressive clinical results with durable complete responses in patients with metastatic melanoma. Recently, the investigators have completed a pilot study treating 6 patients with metastatic ovarian cancer. The TILs are isolated from patients own tumor tissue followed by in vitro expansion and activation for around 4-6 weeks. Before TIL infusion the patients receive 1 week of preconditioning chemotherapy with cyclophosphamide and fludarabine. After TIL infusion Interleukin-2 is administered to support T cell activation and proliferation in vivo.

The investigators recent pilot study has shown TIL therapy in patients with metastatic ovarian cancer to be feasible and tolerable. Mainly transient clinical responses where observed and therefore the investigators plan to combine TIL therapy with checkpoint inhibitors to potentially increase the clinical effect.

DETAILED DESCRIPTION:
Adoptive T cell therapy (ACT) with tumor infiltrating lymphocytes (TIL) has achieved impressive clinical results with durable complete responses in patients with metastatic melanoma. Recently, the investigators have completed a pilot study treating 6 patients with metastatic ovarian cancer. The TILs are isolated from patients own tumor tissue followed by in vitro expansion and activation for around 4-6 weeks. Before TIL infusion the patients receive 1 week of preconditioning chemotherapy with cyclophosphamide and fludarabine. After TIL infusion Interleukin-2 is administered to support T cell activation and proliferation in vivo.

The investigators recent pilot study has shown TIL therapy in patients with metastatic ovarian cancer to be feasible and tolerable. Mainly transient clinical responses where observed and therefore the investigators plan to combine TIL therapy with checkpoint inhibitors to potentially increase the clinical effect.

Objectives:

To evaluate safety and feasibility when treating patients with metastatic ovarian cancer with ACT with TILs in combination with checkpoint inhibitors.

To evaluate treatment related immune responses To evaluate clinical efficacy

Design:

Patients will be screened with a physical exam, medical history, blood samples and ECG.

Patients will be treated with one dose of Ipilimumab 14 days before undergoing surgery to harvest tumor material for TIL production. Patients is admitted on day -8 in order to undergo lymphodepleting chemotherapy with cyclophosphamide and fludara starting day -7. On day -2 patients will start treatment with Nivolumab every 2 weeks for a total of 4 doses to increase the activity of the infused TIL product.

On day 0 patients receive TIL infusion and shortly after starts IL-2 stimulation with a daily subcutaneous dose for a total of 14 days.The patients will followed until progression or up to 5 years.

ELIGIBILITY:
Only patients within the Danish healthcare system are eligible for enrollment.

Inclusion Criteria:

* Histological proven advanced ovarian-, fallopian tube or primary peritoneal cancer with the possibility of surgical removal of tumor tissue of > 1 cm3.
* Progressive or recurrent resistant disease after platin-based chemotherapy (platinum resistant) or progressive or recurrent disease after second line or additional chemotherapy.
* Age: 18 - 70 years.
* ECOG performance status of ≤1 (Appendix 2).
* Life expectancy of > 6 months.
* At least one measurable parameter in accordance with RECIST 1.1 -criteria's.
* No significant toxicities or side effects from previous treatments, except sensoric- and motoric neuropathy and/or alopecia
* Sufficient renal, hepatic and hematological function
* Men and women in the fertile age must use effective contraception. This applies from inclusion and until 6 months after treatment.
* Able to comprehend the information given and willing to sign informed consent

Exclusion Criteria:

* Other malignancies, unless followed for ≥ 5 years with no sign of disease
* Known hypersensitivity to one of the active drugs or one or more of the excipients.
* Severe medical or psychiatric conditions
* Creatinine clearance < 70 ml/min. In selected cases it can be decided to include a patient with a GFR < 70 ml/min with the use of a reduced dose of chemotherapy.
* Acute/chronic infection with HIV, hepatitis, syphilis among others.
* Severe allergies or previous anaphylactic reactions.
* Active autoimmune disease
* Pregnant women and women breastfeeding.
* Need for immunosuppressive treatment e.g. corticosteroids or methotrexate. In selected cases a systemic dose of ≤10 mg prednisolone or a transient planned treatment that can be stopped before TIL therapy can be tolerated.
* Simultaneous treatment with other experimental drugs.
* Simultaneous treatment with other systemic anti-cancer treatments.
* Patients with active and uncontrollable hypercalcaemia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, Prof., M.D., Study Director — Center for Cancer Immune Therapy, Depth of Hematology/Oncology, Copenhagen University Hospital Herlev, Herlev Ringvej 75, DK-2730; Magnus Pedersen, M.D., Principal Investigator — Center for Cancer Immune Therapy, Depth of Hematology/Oncology, Copenhagen University Hospital Herlev, Herlev Ringvej 75, DK-2730
Locations (1):
- Center for Cancer Immune Therapy Dept. of Hematology/oncology, Copenhagen, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- TIL Treated Patients: Ipilimumab Cyclophospamide Fludarabine Nivolumab TILs IL-2
Period: Overall Study
Arm/Group | TIL Treated Patients
Started | 7
All Treated With TILs | 6
Completed | 6
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | TIL Treated Patients
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reported Adverse Events by Type
Description: Determine the safety of TIL therapy in combination with checkpoint inhibitors for patients with ovarian-, fallopian tube or primary peritoneal cancer by reporting adverse events according to CTCAE v. 4.0.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | TIL Treated Patients
Number analyzed (Participants) | 6
Participants
  Performance status drop | 3
  Fatigue | 3
  Nausea | 1
  Vomiting | 1
  Diarrhea | 1
  Hyponatremia | 3
  Infection | 2
  Neutropenia | 6
  Trombocytopenia | 6
  Anemia | 6
  Agammaglobulinemia | 1
  Dyspnea | 1
  Fever | 3
  Colitis | 1
  Dry skin | 1

2. Secondary Outcome: Treatment Related Immune Responses
Description: Ex vivo anti-tumor reactivity of expanded TILs after co-culture measured with flow cytometry.
Time Frame: Until protocol end, until 6 months after TIL infusion
Measure: Count of Participants; unit: Participants
Groups:
- Patient Group: Patients treated with TILs
Arm/Group | Patient Group
Number analyzed (Participants) | 6
Participants | 6

3. Secondary Outcome: Objective Response Rate
Description: Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CAT scan:
  Complete Response (CR) Disappearance of all target lesions (sum of all taget lesions=0) Partial Response (PR) >=30% decrease (vs baseline) of sum of all target lesions dimension Progressive Disease (PD) new lesions or >=20% increase (vs smallest sum of target lesions or nadir) Stable Disease (SD) when sum of all target lesions does not qualify for CR/PR/PD
Time Frame: Assessed up to 12 months after therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | TIL Treated Patients
Number analyzed (Participants) | 6
Participants
  Complete response | 0
  Partial response | 1
  Stabile disease | 5
  Progressive disease | 0

4. Secondary Outcome: Overall Survival
Description: Overall Survival (OS), defined as time from TIL infusion to death
Time Frame: Up to 3 years after TIL infusion
Measure: Median (Full Range); unit: Days
Arm/Group | TIL Treated Patients
Number analyzed (Participants) | 6
Days | 247 [136 to 915]

5. Secondary Outcome: Progression Free Survival
Description: Progression free survival (PFS): Time from TIL infusion to disease progression, relapse or death due to any cause, which ever comes first, will be used as an event.
Time Frame: Up to 12 months after TIL infusion
Measure: Median (Full Range); unit: Days
Arm/Group | TIL Treated Patients
Number analyzed (Participants) | 6
Days | 93 [84 to 342]

ADVERSE EVENTS:
Time Frame: From first therapy and until discontinuation from protocol - up to 12 months after.
Description: Adverse event above grade 2 (CTCAE 4.0)
Arm/Group | TIL Treated Patients
All-Cause Mortality (participants affected / at risk) | 6/6
Serious Adverse Events (participants affected / at risk) | 6/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TIL Treated Patients (N=6)
Colitis (Immune system disorders) | 1 (1) — after ipilimumab
Agammaglobulimia (Blood and lymphatic system disorders) | 1 (1) — B-cell deficiency
Infection (Renal and urinary disorders) | 1 (2) — After TILs and immune suppresion
Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — after TILs
Fatigue (General disorders) | 3 (6)
Nausea (General disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Hyponatremia (Renal and urinary disorders) | 3 (3) — Cyclophosphamide
Neutropenia (Blood and lymphatic system disorders) | 6
Trombocytopenia (Blood and lymphatic system disorders) | 6
Anemia (Blood and lymphatic system disorders) | 6
Fever (General disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIL Treated Patients (N=6)
Vomiting (Gastrointestinal disorders) | 3
nausea (General disorders) | 5
Thyroiditis (Endocrine disorders) | 1 — immune related adverse event
Infection (Infections and infestations) | 2
diarrhea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 2
Oral mucositis (Gastrointestinal disorders) | 3
Obstipation (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Elevated liver enzymes (Hepatobiliary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/74/NCT03287674/Prot_SAP_000.pdf